CLINICAL TRIAL: NCT00921401
Title: Improving the Quality of Asthma Care Using the Internet
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Penn State University (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 662; 5R01HL088590-02 (NIH)
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthma Feedback (Experimental): Each month and before all visits with their asthma care provider, participants will be encouraged to go online and answer a series of questions regarding the types of asthma medications they use and how often they use them, asthma symptoms they have experienced, emergency department visits in the past year, the care they have received for their asthma (e.g., specialist visits) in the past year, and the planned date of their next visit with their asthma care provider. Participants will receive tailored feedback about what questions they should ask their doctor during a subsequent visit, whether or not they should schedule a visit sooner, and links to read more about each recommendation.
  Interventions: Behavioral: Asthma Feedback
- Preventive Feedback (Active Comparator): Each month and before all visits with their primary care provider, participants will be encouraged to go online and answer a series of questions regarding their preventive care. They will receive tailored feedback regarding preventive services, such as pap testing, cancer screenings, and flu shots. Participants will receive tailored feedback regarding preventive services (e.g., cancer screening) that they should discuss with their primary care provider.
  Interventions: Behavioral: Asthma Feedback

INTERVENTIONS:
Behavioral: Asthma Feedback — All participants will log in to the study Web site at least once a month and before all doctor visits. They will answer a series of questions and receive individualized feedback about the types of questions they should ask their doctor.

SUMMARY:
It is important for people with asthma to become involved in their asthma care and management. This study will evaluate an interactive Web site that provides tailored feedback and information to asthma patients and encourages them to ask their doctor specific questions about their asthma care.

DETAILED DESCRIPTION:
Asthma is a common cause of illness and lost productivity, including missed days of work and school, in the United States. It is important for people with asthma to become involved in their treatment and care. Previous studies have shown that encouraging people to ask their doctor for various medical tests and treatments improves preventive care (e.g., cancer screenings), but more research is needed on the effect this can have on asthma management. This study will involve an interactive Web site that will ask patients questions about their asthma symptoms and medications and provide suggestions and feedback on the types of questions patients may want to ask their doctors. By asking questions about their asthma care and increasing communication with their doctor, patients may experience improved quality of asthma care and better asthma control. The purpose of this study is to evaluate the impact of the interactive Web site on asthma control and other measures of asthma management.

This 12-month study will enroll people with asthma. Participants will be randomly assigned to either the Asthma Feedback group or the Preventive Feedback (control) group. Both groups will log in to the study Web site at least once a month for 12 months and before all doctor visits. After logging in to the Web site, participants in the Asthma Feedback group will answer a series of questions about their asthma care. They will then receive information and feedback on the types of questions they should ask their asthma care provider during their next office visit. Participants in the Preventive Feedback group will answer questions and receive information and feedback regarding preventive services (e.g., cancer screening, cholesterol screening) that they should discuss with their primary care provider. At baseline and Months 6 and 12, all participants will complete online questionnaires regarding their asthma and overall health. Study researchers will review participants' medical records and insurance claims data at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Only individuals with persistent asthma will be considered for this study. These definitions are made based on definitions from the National Committee for Quality Assurance (NCQA) and include individuals who meet either criteria A or B:

* A: (Four or more prescription medications used for asthma treatment in 1 year) OR (One or more visits to the emergency room with a principal diagnosis of asthma in 1 year) OR (One or more inpatient hospital visits with a principal diagnosis of asthma in 1 year)
* B: (Four or more outpatient visits with any diagnosis of asthma) AND (two or more claims for a prescription drug used for asthma treatment in 1 year)

Other Inclusion Criteria:

* Speaks and reads English fluently
* Member of Highmark
* Has access to the Internet at home or at work
* Has a valid e-mail address
* No history of more than 20 pack-years of cigarette smoking
* Enrolled in a Highmark health plan offering that includes prescription drug coverage

Exclusion Criteria:

* Does not speak English
* Does not have Internet access at home or work
* Smoked more than 20 pack-years (to exclude possible chronic obstructive pulmonary disease [COPD])
* Does not currently have asthma
* Pregnant
* Unwilling to consent

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 408 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Asthma control - as measured by the Asthma Control Test | Measured at Year 1

SECONDARY OUTCOMES:
Medication adherence, as measured by claims data | Measured at Year 1
Outpatient provider visits, as measured by claims data | Measured at Year 1
Asthma-related emergency department visits, as measured by claims data | Measured at Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Christopher N Sciamanna, MD, MPH, Principal Investigator — Penn State University
Locations (1):
- Penn State Hershey Medical Center, Penn State College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Pool AC, Kraschnewski JL, Poger JM, Smyth J, Stuckey HL, Craig TJ, Lehman EB, Yang C, Sciamanna CN. Impact of online patient reminders to improve asthma care: A randomized controlled trial. PLoS One. 2017 Feb 3;12(2):e0170447. doi: 10.1371/journal.pone.0170447. eCollection 2017. PMID 28158200